CLINICAL TRIAL: NCT05073796
Title: Tonotopische Cochlea-Stimulation Und Der Einfluss Auf Das Vestibularorgan
Brief Title: Cochlear Implant Electrostimulation and the Influence on the Vestibular Organ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Collaborators: Advanced Bionics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 19-062
Record Dates: First submitted 2020-11-27; First posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Deafness Unilateral; Deafness, Bilateral; Deafness Congenital; Deafness, Acquired
Keywords: Deafness, Cochlea Implant
MeSH Terms: conditions — Hearing Loss, Unilateral; Hearing Loss, Bilateral; Deafness | interventions — Cochlear Implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Experimental): Participants will receive the intervention as descibed in the respective section.
  Interventions: Device: Cochlea Implant

INTERVENTIONS:
Device: Cochlea Implant — * examination and documentation of vital signs and concomitant medication
  * application of an cochlea implant loan processor (external body surface) with varying stimulus pattern for vestibular stimulation by means of basal, medial and apical electrodes
  * attraction of an special mask to determine the subjective visual vertical (SVV)
  * assessment of the vertical spatial axis with all electrodes turned off
  * assessment of the vertical spatial axis with all electrodes turned on
  * assessment of the vertical spatial axis while using basal (12-16) and medial (6-11) electrodes
  * assessment of the vertical spatial axis while using basal (12-16) and apical (1-5) electrodes
  * assessment of the vertical spatial axis while using medial (6-11) and apical (1-5) electrodes

SUMMARY:
There is evidence that the sensor function of the utricle in patients with bilateral labyrinthine dysfunction (bilateral vestibulopathy) may improve balance under the influence of high frequency basal stimulation of the cochlea.

The aim of the study is to measure the possible co-stimulation of the utricle (which is determined by the SVV) by tonotopic (frequency-specific) cochlear stimulation and thus to objectify whether the stimulation of the auditory nerve in CI patients also leads to an unavoidable co-stimulation of the vestibular system.

DETAILED DESCRIPTION:
The cochlea is tonotopically structured, i.e. certain frequencies are mapped on a specific part of the cochlea from basal to apical. It is not yet known whether tonotopically differentiated stimulation of the cochlea has an unavoidable side effect on other body systems, such as the vestibular organ. If the labyrinthine dysfunction occurs as a consequence of a CI implantation, this could in the future lead to the possibility of reducing vestibular complications after CI surgery by switching certain electrodes on or off.

In a first investigation phase, a conventional and already implanted CE-certified cochlear implant will be used. The aim of this project is to test certain tonotopic stimulus patterns that stimulate the cochlea by varying the volume within predefined settings. Thus, there is no misuse of the device and no change in performance attributes. Within the framework of the clinical project planned here, the testing of vestibular co-stimulation during normal cochlear stimulation via the basal, medial and apical electrodes of the CI electrode is planned. Under the influence of defined stimulation patterns, the assessment of the subjective visual vertical (SVV) in project participants will be investigated.

The influence of tonotopic stimulation on the SVV result will have a high priority.

ELIGIBILITY:
Inclusion Criteria:

* uni- or bilaterally deafened and deaf patients with cochlear implants (one- or two- sided) from Advanced Bionics (AB), model HiRes 90K and newer
* majority
* given informed consent
* legally competent and mentally able to follow the instructions of the personnel

Exclusion Criteria:

* unsuccessful CI implantation (device or electrode defects, incomplete electrode array insertion, missing neuronal stimulus responses)
* pregnant and/or breastfeeding women
* severe pre- or concomitant disease or reduced general ground condition, so that an outpatient presentation in the ENT polyclinic is not possible
* life expectancy of less than six months
* the patient has received a study medication within the last 30 days within the framework of another study
* simultaneous participation in another clinical intervention study
* anticipated lack of compliance
* alcohol or drug abuse
* the patient is placed in an institution by order of the authorities or court
* patients who are in a dependent or employed relationship with the sponsor, investigator, or their deputy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-01-09 (Actual); Study Completion 2021-01-09 (Actual)

PRIMARY OUTCOMES:
Change of the subjective visual vertical (SVV) with tonotopic CI stimulation | 15 - 30 minutes
  The SVV is determined by wearing a special mask that prevents patients from seeing their spatial position. Instead, they see a light bar in the mask. The head is now tilted to the left and right. After adjusting the body position, the examiner asks to be told when the light bar is perceived to be vertical.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Westhofen, Prof.Dr.med., Principal Investigator — Klinik für Hals- Nasen-Ohrenheilkunde, Uniklinik RWTH Aachen
Locations (1):
- Klinik für Hals-Nasen-Ohrenheilkunde, University Hospital Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nguyen TAK, Cavuscens S, Ranieri M, Schwarz K, Guinand N, van de Berg R, van den Boogert T, Lucieer F, van Hoof M, Guyot JP, Kingma H, Micera S, Perez Fornos A. Characterization of Cochlear, Vestibular and Cochlear-Vestibular Electrically Evoked Compound Action Potentials in Patients with a Vestibulo-Cochlear Implant. Front Neurosci. 2017 Nov 21;11:645. doi: 10.3389/fnins.2017.00645. eCollection 2017. PMID 29209162
- [Background] Bance ML, O'Driscoll M, Giles E, Ramsden RT. Vestibular stimulation by multichannel cochlear implants. Laryngoscope. 1998 Feb;108(2):291-4. doi: 10.1097/00005537-199802000-00025. PMID 9473085
- [Background] Guinand N, Van de Berg R, Cavuscens S, Ranieri M, Schneider E, Lucieer F, Kingma H, Guyot JP, Perez Fornos A. The Video Head Impulse Test to Assess the Efficacy of Vestibular Implants in Humans. Front Neurol. 2017 Nov 14;8:600. doi: 10.3389/fneur.2017.00600. eCollection 2017. PMID 29184530
- [Background] Parkes WJ, Gnanasegaram JJ, Cushing SL, McKnight CL, Papsin BC, Gordon KA. Vestibular evoked myogenic potential testing as an objective measure of vestibular stimulation with cochlear implants. Laryngoscope. 2017 Feb;127(2):E75-E81. doi: 10.1002/lary.26037. Epub 2016 Jun 12. PMID 27291637
- [Background] Jiang D, Cirmirakis D, Demosthenous A. A vestibular prosthesis with highly-isolated parallel multichannel stimulation. IEEE Trans Biomed Circuits Syst. 2015 Feb;9(1):124-37. doi: 10.1109/TBCAS.2014.2323310. Epub 2014 Jul 25. PMID 25073175